CLINICAL TRIAL: NCT03532737
Title: Phase II Non-Randomised Controlled Trial Of Concomitant Immune Check Point Inhibitor With Radiotherapy And Chemotherapy Or Cetuximab In Advanced Non Metastatic Head And Neck Cancer
Brief Title: Concomitant Immune Check Point Inhibitor With Radiochemotherapy in Head And Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuwait Cancer Control Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNIT 01
Record Dates: First submitted 2018-05-06; First posted 2018-05-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Head and Neck Cancer
Keywords: head and neck cancer; check point inhibitor; Pembrolizumab; Chemoradiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Investigational Arm (Experimental): All patients will receive radical chemoradiation in addition to the investigational concomitant check point inhibitor CHEMOTHERAPY: Cisplatin: 100 mg/m2 Q21d D1, D22, D43. OR Cetuximab Loading dose 400 mg/m², one week before radiation then maintenance dose 250 mg/m² weekly, D8, D15, D22, D29, D36, D43.
  PD-1 inhibitor: Pembrolizumab 200 mg administered as an intravenous infusion over 30 minutes every 3 weeks 21 days prior to radiation, then Day 1 of radiation and then every 21 days for total 6 doses
  Intensity modulated radiotherapy (IMRT) techniques will be used. A total dose of 66-70 Gy/ 30-35 Fr over 6-7 weeks will be delivered to the primary site and draining lymphatics using simultaneous Integrated Boost (SIB).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Adding PD-1 inhibitor to the standard of care
  Other Names: Keytruda

SUMMARY:
Background: Locally advanced head and neck cancer (HNC) is a challenge as, in spite of initial good control with chemoradiation, the majority of patients fails systemically. In the last 2 years, immune check points inhibitors (mainly Programmed Death (PD)-1 inhibitors) were approved for metastatic/recurrent HNC. The favorable toxicity profile and durable responses was the main benefit of these drugs along the scope of cancers they were approved for.

Aim of the study and methods: This will be a phase II non-randomized trial to define safety and efficacy of combining the PD-1 inhibitor pembrolizumab given concomitantly with the usual standard of care chemoradiation/bioradiation for locally advanced non-nasopharyngeal HNC. Primary end point will be assessment of toxicity and tolerability while the secondary end points will be response rates (RR) and progression free survival (PFS)

DETAILED DESCRIPTION:
Among the Gulf Countries Collaboration Council (GCCC) states, HNC account for 11.5 per 100,000 population. The incidence of HNC in Kuwait is 3.8 per 100,000 population. This, as an example, accounts for about 12.7% of all cancer cases during the period from 1993 to 1999.

Rationale of Immunotherapy in Head and Neck Cancers Cancer immunotherapy principle is functional restoration of certain signaling pathways of the immune system. These pathways help to counteract different tumour evasion strategies. These may include reduced antigen processing and presentation, increased tumour-permissive cytokine profiles, creating an immunosuppressive microenvironment, cellular immune escape, and induction of non-functioning T-cells either by an increase of co-inhibitory receptors; e.g. cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) or PD-1 or decreased co-stimulatory receptors. , Immune checkpoints pathway is the most studied so far. It works by regulating the duration and extent of immune system activity through negative feedback signals. These include CTLA-4, PD-1 and PD-L1/PD-L2.

Head and neck cancers use different immune evasion mechanisms. Immune dysfunction has been implicated in carcinogenesis of human papillomavirus (HPV)-positive oropharyngeal cancer as well as cases linked to smoking.

PD-1 and PD-L1 interplay is extremely interesting. A French group from Sorbonne attempted to explain the better prognosis of HPV-positive tumours of the oropharynx. They examined PD-1 and PD-L1 expression in 64 cases, mostly of oropharyngeal origin. Infiltration of PD-1+ T-lymphocytes was a favourable prognostic factor in HPV-related disease. This also was confirmed by others, where expression of PD-L1 is common regardless of HPV status.

Safety Issues At the University of Pennsylvania, safety of ipilimumab with hypofractionated palliative radiotherapy (RT) was tested in a phase I study. There was no grade 4 or higher toxicities in the cohort of 21 patients. The most common grade 3 toxicity was anemia, that is unlikely to be related to the RT.

Anti-PD-1 agents have a better safety profile than anti-CTLA4 agents. The rate of grade 3 toxicity for pembrolizumab in NSCLC in KEYNOTE-001 was <10%, including a 1.8% rate of grade 3 pneumonitis. And in modern stereotactic body radiotherapy (SBRT) series, the rate of grade 3 radiation pneumonitis is <5%.

Interaction between Immunotherapy and Chemotherapy Classical speaking, chemotherapy (CTH) is very immune suppressive and therefore not an ideal partner for combining with vaccines (and of course other types of immunotherapy), that require an active response. Analysis of the potential interaction of CTH and immunotherapy reveals that there are many mechanisms of synergy. This suggests that the optimal treatment of cancer may include combination of immunotherapy-CTH in an optimal sequential manner.

These mechanism may include the synergistic effect of CTH in reducing tumor load and shedding antigens, as well as the inhibitory effect on regulatory cells and myeloid suppressive cells. On the other way around, immunotherapy can markedly enhance the response to CTH by activating the immune response prior to antigen release, as well as expanding activated T cells that have seen the tumor antigen.

In 2016, Langer et al published their work in the KEYNOTE-021 of combining carboplatin/pemetrexed with pembrolizumab. The combination of the chemotherapy with immunotherapy in advanced NSCLC showed tolerability as well as effectiveness. This lead to the approval of this combination in May 2017 by FDA.

Ongoing Concomitant Immunotherapy and Radiotherapy Trials in HNC Four ongoing studies are explore inhibition of the PD-1/PD-L1 in combination with definitive RT with or without cisplatin or cetuximab. These are trial: NCT02707588 assessing safety of pembrolizumab vs cetuximab in combination with radiation in non-platinum eligible patients. NCT03040999 (KEYNOTE-412) design added pembrolizumab to chemotherapy with post radiation consolidation as compared to platinum-radiation. NCT02999087 is comparing the combination of avelumab-cetuximab-radiation to cetuximab-radiation or cisplatin-radiation (REACH Trial). NCT02952586 (JAVELIN trail) is testing combination of avelumab with standard of care. RTOG 3504 examines the efficacy and safety of nivolumab in the definitive and adjuvant settings (NCT02764593). Finally, IRX-2 (citoplurikin), a primary human cell-derived biologic with multiple active cytokine components, is being tested in a randomized phase II trial of neoadjuvant and adjuvant therapy in patients with newly diagnosed curative resectable stages II, III, or IVA oral cavity cancer (NCT02609386).

Gaps in Design of ongoing Trials However, most of the studies testing the value of addition of immunotherapy to standard of care, are designed to continue immunotherapy for 4-12 months after finishing radical chemoradiation. This, in our opinion, will give mixed results and affect the conclusion of the survival benefit if found. Extrapolated from many adjuvant clinical trials, the disease control can be attributed to the length of the whole duration of treatment rather than the specific agent used. Moreover, there is no definite duration of this adjuvant immunotherapy in the ongoing trials i.e. they give a wide range of cycles and time. For example, the recruiting KEYNOTE-412 designed for 14 cycles of pembrolizumab while RTOG 3504 will try to give 7 adjuvant cycles (will be determined based on first 8 patients tolerance).

Another point in these trials design; although designed to be multicentric, most of recruiting centers are located in Europe and USA. This will limit the validity of the data and results when other countries (especially in Asia) try to adopt the treatment protocols. Based on many published data, the HNC in Eastern countries and among Asian showed different clinical and biological characteristics e.g. mostly HPV negative, related to tobacco chewing and poor nutritional status.

Lastly, the ongoing trial for nivolumab with RT in locally advanced head and neck cancer (LAHNC) is assessing the safety and efficacy. However, pembrolizumab has already published its phase Ib data extended from the large cohort of many solid tumors. In contrary, avelumab has no published supporting data (so far) regarding this indication from phase II trials. They depend largely upon their safety profiles from the pooled previous studies and/or the other subsites of diseases. As mentioned earlier, there is ongoing NCT02707588 Trial is assessing pembrolizumab safety with radiation vs cetuximab-radiation in cisplatin non-eligible patients.In the current trial, we are trying to fill this gap by testing the efficacy and safety of pembrolizumab with radical chemoradiation in all cases of LAHNC.

Post-Treatment Evaluations Post-treatment evaluations will start 4 weeks after completion of radiation therapy. The 4th week post-treatment evaluations will consist of a physical examination, hematology and biochemistry profiles, tumor assessments (by palpation) and an objective assessment of adverse events which may have occurred since completing treatment. Radiological assessment of response will be done 8-10 weeks post treatment. Responses will be reported according to irRECIST criteria.

Subsequent Follow-up evaluations will commence after the 8 week post-treatment, every four weeks (±1 week) for years one and every 8 weeks for year two, and then, every 4 months (± 2 weeks) for year three to five. The evaluations in the first year will consist of a physical examination, hematology and chemistry profiles, Quality of Life, imaging/diagnostic assessments, and tumor assessments. Evaluations in year 2-5 will consist of a physical examination, imaging/diagnostic, and tumor assessments.

Statistical methods and consideration.

* Statistical package for social sciences (SPSS) version 16. Quantitative variables will be summarized using mean and standard deviation (SD), median minimum and maximum values. Qualitative data will be summarized using frequencies and percentage.
* Overall survival will be calculated from the date of histological diagnosis.
* Progression free survival (PFS) will be calculated from the date of starting of treatment till disease progression and death whichever comes first.
* Survival analysis will be done using Kaplan- Meier, comparisons will be done using Log-rank test.
* Differences will be considered significant when p was 0.05 and highly significant when p 0.01.
* Patients lost for follow up with disease will be considered as dead.
* At the time of data analysis stratification of the patients according to sub sites, prognostic and risk factors including HPV status will be done.

ELIGIBILITY:
Inclusion Criteria:

* The patient has pathologically proven squamous cell carcinoma arising in the oropharynx, hypopharynx, oral cavity, or larynx
* The patient has stage III or IVA disease with an expected survival of 12 months.
* The patient is medically suitable to withstand a course of definitive radiation therapy & chemotherapy.
* Karnofsky performance status is > 60.
* The patient must have achieved lawful age to provide informed consent according to local or national law .
* Laboratory values performed within 14 days prior to concurrent chemotherapy should be as follows:

  i) Absolute neutrophil count (ANC) ≥ 2000/mm ii) Platelet count ≥ 100.000/mm iii) Hemoglobin ≥ 10g/dl or 100g/L iv) Urea and serum creatinine ≤ 1.5 mg/dl. (for cisplatin) v) Creatinine clearance ≥ 50 ml/min. (for cisplatin) vi) serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT) ≤ 2 × upper limit of laboratory normal vii) Serum calcium within normal limits.
* Has provided tissue for Programmed Cell Death Receptor Ligand 1 (PD-L1) biomarker analysis from a core or excisional biopsy
* Has evaluable tumor burden (measurable and/or non-measurable tumor lesions) assessed by computed tomography scan or magnetic resonance imaging, based on RECIST version 1.1
* Is eligible for definitive chemoradiation (CRT) and not considered for primary surgery based on investigator decision
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study therapy
* Female and male participants of reproductive potential must agree to use adequate contraception throughout the study period and for up to 180 days after the last dose of study therapy

Exclusion Criteria:

* The patient has evidence of distant metastatic disease.
* The patient has received prior systemic chemotherapy within the last three years.
* The patient has undergone previous surgery for the tumor, other than biopsy.
* The patient has received prior radiation therapy to the H&N.
* The patient's radiation therapy is considered to be a part of a postoperative regimen following primary surgical resection.
* The patient is pregnant or breast feeding.
* The patient has a medical (e.g. renal impairment) or psychological condition that would not permit the patient to complete the trial or sign informed consent.
* Has received prior therapy with an anti-Programmed Cell Death Receptor 1 (PD-1), anti-PD-L1, anti-Programmed Cell Death Receptor Ligand 2 (PD-L2) agent or with an agent directed to another co-inhibitory T-cell receptor or has previously participated in clinical studies with immunotherapy
* Has received a live vaccine within 30 days prior to the first dose of study therapy
* Has not recovered from major surgery prior to starting study therapy
* Has known active Hepatitis B or C
* Has known history of Human Immunodeficiency Virus (HIV)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study therapy
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment.
* Has history of a diagnosed and/or treated hematologic or primary solid tumor malignancy, unless in remission for at least 5 years prior to randomization
* Has had previous allogeneic tissue/solid organ transplant
* Has active infection requiring systemic therapy
* Has a history of severe hypersensitivity reaction to Pembrolizumab, Cisplatin, cetuximab or radiotherapy or their analogs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | From the first dose of pembrolizumab to 28 days after the completion of radiation therapy
  A pembrolizumab attributable, dose-limiting toxicity (DLT) will be defined as follows:
  1) Any ≥ grade 3 adverse event (CTCAE, v. 4) that is related to pembrolizumab that does not resolve to grade 1 or less within 28 days; 2) A delay in radiotherapy of > 2 weeks due to toxicity related to pembrolizumab; 3) Inability to complete radiotherapy due to toxicity related to pembrolizumab; 4) Inability to receive an adequate dose (≥ 70%) of cisplatin or cetuximab due to toxicity definitely related to pembrolizumab.
Response Rate | 3 years
  Response rates according to irRECIST criteria

SECONDARY OUTCOMES:
Locoregional control rates | 5 years
  Number of local disease progression events
Progression free survival | 5 years
  Number of local or distant disease progression events
Overall survival | 5 years initially (longer follow up will be done)
  Number of cancer-related deaths

OTHER OUTCOMES:
Patients' Quality of life (QoL) | 5 years initially
  QoL assessment by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa S El-Sherify, MD, Principal Investigator — Kuwait Cancer Control Center
Locations (1):
- Kuwait Cancer Control Center, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Kuwait Cancer Registry: Annual Report 2013. Ministry of Health Publications
- [Background] Thompson LDR. Squamous cell carcinoma variants of the head and neck. Current Diagnostic Pathology (2003) 9, 384 -396
- [Background] Vokes EE, Weichselbaum RR, Lippman SM, Hong WK. Head and neck cancer. N Engl J Med. 1993 Jan 21;328(3):184-94. doi: 10.1056/NEJM199301213280306. No abstract available. PMID 8417385
- [Background] Carvalho AL, Nishimoto IN, Califano JA, Kowalski LP. Trends in incidence and prognosis for head and neck cancer in the United States: a site-specific analysis of the SEER database. Int J Cancer. 2005 May 1;114(5):806-16. doi: 10.1002/ijc.20740. PMID 15609302
- [Background] Pignon JP, le Maitre A, Maillard E, Bourhis J; MACH-NC Collaborative Group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): an update on 93 randomised trials and 17,346 patients. Radiother Oncol. 2009 Jul;92(1):4-14. doi: 10.1016/j.radonc.2009.04.014. Epub 2009 May 14. PMID 19446902
- [Background] Bernier J, Cooper JS, Pajak TF, van Glabbeke M, Bourhis J, Forastiere A, Ozsahin EM, Jacobs JR, Jassem J, Ang KK, Lefebvre JL. Defining risk levels in locally advanced head and neck cancers: a comparative analysis of concurrent postoperative radiation plus chemotherapy trials of the EORTC (#22931) and RTOG (# 9501). Head Neck. 2005 Oct;27(10):843-50. doi: 10.1002/hed.20279. PMID 16161069
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Kimura H, Sakai K, Arao T, Shimoyama T, Tamura T, Nishio K. Antibody-dependent cellular cytotoxicity of cetuximab against tumor cells with wild-type or mutant epidermal growth factor receptor. Cancer Sci. 2007 Aug;98(8):1275-80. doi: 10.1111/j.1349-7006.2007.00510.x. Epub 2007 May 13. PMID 17498200
- [Background] Yang X, Zhang X, Mortenson ED, Radkevich-Brown O, Wang Y, Fu YX. Cetuximab-mediated tumor regression depends on innate and adaptive immune responses. Mol Ther. 2013 Jan;21(1):91-100. doi: 10.1038/mt.2012.184. Epub 2012 Sep 18. PMID 22990672
- [Background] Lattanzio L, Denaro N, Vivenza D, Varamo C, Strola G, Fortunato M, Chamorey E, Comino A, Monteverde M, Lo Nigro C, Milano G, Merlano M. Elevated basal antibody-dependent cell-mediated cytotoxicity (ADCC) and high epidermal growth factor receptor (EGFR) expression predict favourable outcome in patients with locally advanced head and neck cancer treated with cetuximab and radiotherapy. Cancer Immunol Immunother. 2017 May;66(5):573-579. doi: 10.1007/s00262-017-1960-8. Epub 2017 Feb 14. PMID 28197666
- [Background] Allen CT, Clavijo PE, Van Waes C, Chen Z. Anti-Tumor Immunity in Head and Neck Cancer: Understanding the Evidence, How Tumors Escape and Immunotherapeutic Approaches. Cancers (Basel). 2015 Dec 9;7(4):2397-414. doi: 10.3390/cancers7040900. PMID 26690220
- [Background] Ferris RL. Immunology and Immunotherapy of Head and Neck Cancer. J Clin Oncol. 2015 Oct 10;33(29):3293-304. doi: 10.1200/JCO.2015.61.1509. Epub 2015 Sep 8. PMID 26351330
- [Background] Tommasino M. The human papillomavirus family and its role in carcinogenesis. Semin Cancer Biol. 2014 Jun;26:13-21. doi: 10.1016/j.semcancer.2013.11.002. Epub 2013 Dec 4. PMID 24316445
- [Background] Badoual C, Hans S, Merillon N, Van Ryswick C, Ravel P, Benhamouda N, Levionnois E, Nizard M, Si-Mohamed A, Besnier N, Gey A, Rotem-Yehudar R, Pere H, Tran T, Guerin CL, Chauvat A, Dransart E, Alanio C, Albert S, Barry B, Sandoval F, Quintin-Colonna F, Bruneval P, Fridman WH, Lemoine FM, Oudard S, Johannes L, Olive D, Brasnu D, Tartour E. PD-1-expressing tumor-infiltrating T cells are a favorable prognostic biomarker in HPV-associated head and neck cancer. Cancer Res. 2013 Jan 1;73(1):128-38. doi: 10.1158/0008-5472.CAN-12-2606. Epub 2012 Nov 7. PMID 23135914
- [Background] Lin Z, Xu Y, Zhang Y, He Q, Zhang J, He J, Liang W. The prevalence and clinicopathological features of programmed death-ligand 1 (PD-L1) expression: a pooled analysis of literatures. Oncotarget. 2016 Mar 22;7(12):15033-46. doi: 10.18632/oncotarget.7590. PMID 26930715
- [Background] Seiwert TY, Burtness B, Mehra R, Weiss J, Berger R, Eder JP, Heath K, McClanahan T, Lunceford J, Gause C, Cheng JD, Chow LQ. Safety and clinical activity of pembrolizumab for treatment of recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-012): an open-label, multicentre, phase 1b trial. Lancet Oncol. 2016 Jul;17(7):956-965. doi: 10.1016/S1470-2045(16)30066-3. Epub 2016 May 27. PMID 27247226
- [Background] Chow LQM, Haddad R, Gupta S, Mahipal A, Mehra R, Tahara M, Berger R, Eder JP, Burtness B, Lee SH, Keam B, Kang H, Muro K, Weiss J, Geva R, Lin CC, Chung HC, Meister A, Dolled-Filhart M, Pathiraja K, Cheng JD, Seiwert TY. Antitumor Activity of Pembrolizumab in Biomarker-Unselected Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma: Results From the Phase Ib KEYNOTE-012 Expansion Cohort. J Clin Oncol. 2016 Nov 10;34(32):3838-3845. doi: 10.1200/JCO.2016.68.1478. Epub 2016 Sep 30. PMID 27646946
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Ehlers G, Fridman M. Abscopal effect of radiation in papillary adenocarcinoma. Br J Radiol. 1973 Mar;46(543):220-2. doi: 10.1259/0007-1285-46-543-220. No abstract available. PMID 4706791
- [Background] Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, Kitano S, Mu Z, Rasalan T, Adamow M, Ritter E, Sedrak C, Jungbluth AA, Chua R, Yang AS, Roman RA, Rosner S, Benson B, Allison JP, Lesokhin AM, Gnjatic S, Wolchok JD. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31. doi: 10.1056/NEJMoa1112824. PMID 22397654
- [Background] Kalbasi A, June CH, Haas N, Vapiwala N. Radiation and immunotherapy: a synergistic combination. J Clin Invest. 2013 Jul;123(7):2756-63. doi: 10.1172/JCI69219. Epub 2013 Jul 1. PMID 23863633
- [Background] Demaria S, Golden EB, Formenti SC. Role of Local Radiation Therapy in Cancer Immunotherapy. JAMA Oncol. 2015 Dec;1(9):1325-32. doi: 10.1001/jamaoncol.2015.2756. PMID 26270858
- [Background] Schaue D, McBride WH. Opportunities and challenges of radiotherapy for treating cancer. Nat Rev Clin Oncol. 2015 Sep;12(9):527-40. doi: 10.1038/nrclinonc.2015.120. Epub 2015 Jun 30. PMID 26122185
- [Background] Szturz P, Vermorken JB. Immunotherapy in head and neck cancer: aiming at EXTREME precision. BMC Med. 2017 Jun 2;15(1):110. doi: 10.1186/s12916-017-0879-4. PMID 28571578
- [Background] Theurich S, Rothschild SI, Hoffmann M, Fabri M, Sommer A, Garcia-Marquez M, Thelen M, Schill C, Merki R, Schmid T, Koeberle D, Zippelius A, Baues C, Mauch C, Tigges C, Kreuter A, Borggrefe J, von Bergwelt-Baildon M, Schlaak M. Local Tumor Treatment in Combination with Systemic Ipilimumab Immunotherapy Prolongs Overall Survival in Patients with Advanced Malignant Melanoma. Cancer Immunol Res. 2016 Sep 2;4(9):744-54. doi: 10.1158/2326-6066.CIR-15-0156. Epub 2016 Jul 27. PMID 27466265
- [Background] Tang C, Welsh JW, de Groot P, Massarelli E, Chang JY, Hess KR, Basu S, Curran MA, Cabanillas ME, Subbiah V, Fu S, Tsimberidou AM, Karp D, Gomez DR, Diab A, Komaki R, Heymach JV, Sharma P, Naing A, Hong DS. Ipilimumab with Stereotactic Ablative Radiation Therapy: Phase I Results and Immunologic Correlates from Peripheral T Cells. Clin Cancer Res. 2017 Mar 15;23(6):1388-1396. doi: 10.1158/1078-0432.CCR-16-1432. Epub 2016 Sep 20. PMID 27649551
- [Background] Zhao J, Yorke ED, Li L, Kavanagh BD, Li XA, Das S, Miften M, Rimner A, Campbell J, Xue J, Jackson A, Grimm J, Milano MT, Spring Kong FM. Simple Factors Associated With Radiation-Induced Lung Toxicity After Stereotactic Body Radiation Therapy of the Thorax: A Pooled Analysis of 88 Studies. Int J Radiat Oncol Biol Phys. 2016 Aug 1;95(5):1357-1366. doi: 10.1016/j.ijrobp.2016.03.024. Epub 2016 Mar 25. PMID 27325482
- [Background] Lake RA, Robinson BW. Immunotherapy and chemotherapy--a practical partnership. Nat Rev Cancer. 2005 May;5(5):397-405. doi: 10.1038/nrc1613. PMID 15864281
- [Background] Langer CJ, Gadgeel SM, Borghaei H, Papadimitrakopoulou VA, Patnaik A, Powell SF, Gentzler RD, Martins RG, Stevenson JP, Jalal SI, Panwalkar A, Yang JC, Gubens M, Sequist LV, Awad MM, Fiore J, Ge Y, Raftopoulos H, Gandhi L; KEYNOTE-021 investigators. Carboplatin and pemetrexed with or without pembrolizumab for advanced, non-squamous non-small-cell lung cancer: a randomised, phase 2 cohort of the open-label KEYNOTE-021 study. Lancet Oncol. 2016 Nov;17(11):1497-1508. doi: 10.1016/S1470-2045(16)30498-3. Epub 2016 Oct 10. PMID 27745820
- [Background] Mehanna H, Franklin N, Compton N, Robinson M, Powell N, Biswas-Baldwin N, Paleri V, Hartley A, Fresco L, Al-Booz H, Junor E, El-Hariry I, Roberts S, Harrington K, Ang KK, Dunn J, Woodman C. Geographic variation in human papillomavirus-related oropharyngeal cancer: Data from 4 multinational randomized trials. Head Neck. 2016 Apr;38 Suppl 1(Suppl 1):E1863-9. doi: 10.1002/hed.24336. Epub 2016 Jan 8. PMID 26749143
- See also: Cancer Research UK. Accessed [January] [2018] — http://cancerresearchuk.org/health-professional/cancer-statistics/statistics-by-cancer-type/oral-cancer/incidence
- See also: Kulkarni MR. Head and neck cancer Burden in India. Internat J of Head and Neck Surg. 2013; 4 (1): 29-35 — https://pdfs.semanticscholar.org/406e/5fbbcb95c8be01adc0e9771c613ecbee7baf.pdf
- See also: The Gulf Federation for Cancer Control Guidelines. Last Accessed August 2020 — https://gffcc.org/home/wp-content/uploads/2016/10/images_GFFCC_Guidelines_Part-2.pdf
- See also: NCCN Clinical Practice Guidelines in Oncology. Head and Neck. In NCCN Guidelines, Version 1.2018 Edition 2018 — https://www.nccn.org/professionals/physician_gls/pdf/head-and-neck.pdf
- See also: Clinical Trials Protocols. Accessed Feb 2018 — https://clinicaltrials.gov/ct2/show/NCT02707588.
- See also: Clinical Trials Protocols. Accessed Feb 2018 — https://clinicaltrials.gov/ct2/show/study/NCT03040999.
- See also: Clinical Trials Protocols. Accessed Feb 2018 — https://clinicaltrials.gov/ct2/show/NCT02999087.
- See also: Clinical Trials Protocols. Accessed Feb 2018 — https://clinicaltrials.gov/ct2/show/NCT02952586.
- See also: Clinical Trials Protocols. Accessed Feb 2018 — https://clinicaltrials.gov/ct2/show/NCT02764593.
- See also: Clinical Trials Protocols. Accessed Feb 2018 — https://clinicaltrials.gov/ct2/show/NCT02609386.